CLINICAL TRIAL: NCT05496855
Title: Can Machine Learning and Patient-reported Outcomes be Used in Remote Care in People With Rheumatic Diseases
Brief Title: Remote Care in People With Rheumatoid Arthritis
Acronym: NOR-Flare
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Diakonhjemmet Hospital (Other)
Responsible Party: Principal Investigator, Anne Therese Tveter, Principal Investigator, Senior researcher/Assosiate Professor, Diakonhjemmet Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REK 457358
Record Dates: First submitted 2022-08-04; First posted 2022-08-11 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Rheumatoid Arthritis
Keywords: remote care
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Control Groups; Remote Patient Monitoring

STUDY DESIGN:
Intervention Model Description: Randomized controlled non-inferiority trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Conventional follow-up (Active Comparator): Conventional follow-up strategy with blood tests and face-to-face visits at the hospital every 6 months
  Interventions: Other: Conventional follow-up
- Remote monitoring (Experimental): Monthly remote monitoring of patient-reported outcomes and triage of patients using an algorithm will guide healthcare providers in scheduling patients for a video consultation or face-to-face hospital visits.
  Interventions: Other: Remote monitoring

INTERVENTIONS:
Other: Conventional follow-up — Patients in the conventional/usual care arm will be treated according to current conventional follow-up regimen with PROs, blood tests, and face-to-face visits with an experienced nurse or a rheumatologist every 6 months. They can contact the hospital if they are experience worsening of their disease.
  Other Names: Control group
  Arms: Conventional follow-up
Other: Remote monitoring — The patients in the remote monitoring arm will use a web-app (Youwell) for self-reporting patient reported outcomes (PROs) and CRP/ESR, displaying results for PROs over time, and for synchronous (video) or asynchronous (chat) communication with healthcare providers. The patients will receive a SMS reminder for "tasks" (e.g., self-reporting PROs or registering results from blood tests) every month.
  A study coordinator/nurse will monitor the PROs and blood test (CRP/ESR) results, and respond to chat messages. Based on the algorithm, a triaging functionality in the Youwell platform will aid healthcare providers in highlighting which patients needs attention.
  Other Names: Intervention group
  Arms: Remote monitoring

SUMMARY:
This study is a 24-months, non-inferiority randomized, controlled trial with two parallel arms to determine if a new follow-up strategy for patients with RA is non-inferior in maintaining comprehensive disease control measured as simultaneous maintenance of structural, functional and clinical treatment target at 2-year follow-up compared to the conventional follow-up regimen with regular hospital visits.

DETAILED DESCRIPTION:
The study will include Norwegian adult males and females with rheumatoid arthritis. Eligible patients that consent to participation will be randomized to two groups:

* Control group: conventional follow-up strategy with blood tests, patient-reported outcomes (PROs), and pre-scheduled visits at the hospital every 6th month.
* Remote monitoring: monthly remote monitoring of PROs and triage of patients using an algorithm will guide healthcare providers in scheduling patients for a video consultation or face-to-face hospital visits.

Participants will be followed for 24 months. Primary outcome is proportionn maintaining comprehensive disease control measured as simultaneous maintenance of structural, functional and clinical treatment target at 2-year follow-up1.

* Structural: Assessed with radiographs of hands and feet according to the van der Heijde modified Sharpe score (subscores for erosions (0-280) and joint space narrowing (0-168)), with a total range of 0-448. Maintenance of structural treatment target is defined as change in total score <1 unit/year (<2 units from inclusion to 2-year follow-up).
* Functional: Measured by Modified Health Assessment Questionnaire (MHAQ) measured on a scale from 0.00 to 3.00, where a change of 0.25 is considered clinical important3. Maintenance of functional treatment target is defined as a worsening <0.25 from inclusion to 2-year follow-up.
* Clinical: Measured by DAS28, categorized into remission (<2.6), low disease activity (2.6 to ≤3.2), moderate disease activity (3.2 to ≤5.1) and high disease activity (>5.1). Maintenance of clinical treatment target is defined disease activity category at 2-year follow-up ≤ baseline category.

We will use a 15% non-inferiority margin.

The study will comprise an internal pilot study the first 6 months for all participants in the intervention group.

The study will also include qualitative research including semi-structured interviews and observations of patients in the intervention group and health professionals involved in the study. The interviews will explore experiences with remote monitoring and video consultations.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant, non-nursing female ≥18 years of age at screening
* Patients with a diagnosis of RA who fulfil the 2010 ACR/EULAR diagnostic criteria24 (see Appendix 5, 10.4)
* Medical treatment with cs/ts/bDMARDs (incl. prednisolone) considered stable by the healthcare provider the last 6 months
* Low disease activity or remission (CDAI<10 / DAS28<3.2) at inclusion
* <2 swollen joints
* Not deemed inappropriate for remote monitoring by the healthcare provider
* Capable of understanding and signing an informed consent form
* Access to a smartphone or tablet
* Able to speak and understand Norwegian language

Exclusion Criteria:

Medical conditions:

* Major co-morbidities, such as severe malignancies, severe diabetes mellitus, severe infections, uncontrollable hypertension, severe cardiovascular disease (NYHA class III or IV), severe respiratory diseases, and/or cirrhosis.
* Indications of active tuberculosis (TB)
* Treated with intravenous DMARD (e.g., rituximab and infliximab)

Diagnostic assessments:

* Abnormal renal function, defined as serum creatinine >142 µmol/L in female and >168 µmol/L in male, or glomerular filtration rate (GFR) <40 mL/min/1.73 m2
* Abnormal liver function (defined as Aspartate Transaminate (AST)/Alanine Transaminase (ALT) >3 x upper normal limit), active or recent hepatitis
* Leukopenia and/or thrombocytopenia

Other:

* Pregnancy and/or breastfeeding (current at screening or planned within the duration of the study)
* Severe psychiatric or mental disorders, alcohol abuse or other substance abuse, language barriers or other factors which makes adherence to the study protocol impossible.
* Deemed unsuitable for remote monitoring by medical doctor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 228 (Estimated)
Dates: Start 2022-09-29 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2028-10-14 (Estimated)

PRIMARY OUTCOMES:
Proportion maintaining comprehensive disease control | Baseline and 2 years
  Comprehensive disease control measured as simultaneous maintenance of structural, functional and clinical treatment target at 2-year follow-up.
  * Structural: Radiographs of hands and feet according to the van der Heijde modified Sharpe score, with a total range of 0-448. Maintenance of structural treatment target is defined as change in total score <1 unit/year (<2 units from inclusion to 2-year follow-up).
  * Functional: Modified Health Assessment Questionnaire (MHAQ) measured on a scale from 0.00 to 3.00, where a change of 0.25 is considered clinical important. Maintenance of functional treatment target is defined as a worsening <0.25 from inclusion to 2-year follow-up.
  * Clinical: DAS28, categorized into remission (<2.6), low disease activity (2.6 to ≤3.2), moderate disease activity (3.2 to ≤5.1) and high disease activity (>5.1). Maintenance of clinical treatment target is defined disease activity category at 2-year follow-up ≤ baseline category.

SECONDARY OUTCOMES:
Change in joint damage progression | Baseline and 2 years
  Joint damage progression from inclusion to 2-year follow-up assessed with radiographs of hands and feet according to the van der Heijde modified Sharpe score (subscores for erosions (0-280) and joint space narrowing (0-168)), with a total range of 0-448. Measured as a continuous variable.
Self-reported disease activity (intervention group) | Monthly until 2 years
  Measured with patient global assessment of disease activity (0-10 scale, 0=no disease activity), estimated as change across all timepoints
Self-reported disease activity (control group) | Baseline, 6 months, 12 months, 18 months and 2 years
  Measured with patient global assessment of disease activity (0-10 scale, 0=no disease activity), estimated as change across all timepoints
Health-related quality of life | Baseline, 6 months, 12 months, 18 months and 2 years
  Measured with EQ5D-5L, 5 questions used to calculate an utility score (0-1, 1= best health), assessed as a total score across all timepoints
Proportion in remission/low disease activity (CDAI) | Baseline and 2 years
  Measured with CDAI (patient global assessment of disease activity, number of tender and swollen joints, physician assessment of disease activity). Remission/low disease activity defined as CDAI <10.
Proportion in remission/low disease activity (DAS28) | Baseline and 2 years
  Measured with DAS28 (patient global assessment of disease activity, CRP/ESR, number of tender and swollen joints). Remission/low disease activity defined as DAS28 <3.2.
Disease activity in conjunction with consultation (DAS28) | Any consultation from baseline to 2 years
  Measured with DAS28 (patient global assessment of disease activity, CRP/ESR, number of tender and swollen joints).
  DAS28 score: <2.6= remission; 2.6-<3.2=low disease activity; 3.2 -5.1= moderate disease activity; >5.2= high disease activity
Disease activity in conjunction with consultation (CDAI) | Any consultation from baseline to 2 years
  Measured with CDAI (patient global assessment of disease activity, number of tender and swollen joints, physician assessment of disease activity).
  CDAI score: <=2.8 = remission; >2.8 - <=10 = low disease activity; >10 - <=22 = moderate disease activity; >22 = high disease activity
Health care utilization | Baseline, 6 months, 12 months, 18 months, 2 years
  Costs related to self-reported healthcare use in primary and secondary health care. Patients will be asked if they have been seeking healthcare (yes/no), if yes, they will be asked to specify type of healthcare use and time used. This information will also be collected from national register data.
Patient-reported disease flares (intervention group) | Every month until 2 years
  Patient-reported experience of a significant worsening of symptoms (reflecting a flare in disease activity), response options: no, yes, uncertain. If yes or uncertain, they will be asked which date the flare occurred and the number of days it lasted.
Patient-reported disease flares (control group) | 6 months, 12 months, 18 months, 2 years
  Patient-reported experience of a significant worsening of symptoms (reflecting a flare in disease activity), response options: no, yes, uncertain. If yes or uncertain, they will be asked which date the flare occurred and the number of days it lasted.
Adverse events | Through study completion, maximum 2 years
  Number of adverse events, serious adverse events, and withdrawals because of adverse events.
Number of consultations/contacts at the hospital | From baseline to 2 years
  Reported by research nurse or study doctor when in contact with a patient.
Activity impairment (intervention group) | Baseline and monthly until 2 years
  Item no.6 from Work Productivity and Activity Impairment (WPAI): self-reported activity impairment on a NRS 0-10; higher value indicate worse outcome.
Activity impairment (control group) | Baseline, 6 months, 12 months, 18 months, 2 years
  Item no.6 from Work Productivity and Activity Impairment (WPAI): self-reported activity impairment on a NRS 0-10; higher value indicate worse outcome.
Costs related to hospital visits | Baseline
  Self-reported travel distance (km and time) and way of transport (walking, bicycle, privat car, public transportation, taxi, airplane, other) in conjunction with consultation at the hospital
The need to take time off for hospital visits or video consultation | Baseline
  If in paid work, the need to take time off from work is indicated as yes or no.
C-Reactive Protein (CRP) (intervention group) | Baseline, 3, 6, 9, 12, 15, 18, 21 months and 2 years
  Blood test at hospital or general practitioner
C-Reactive Protein (CRP) (control group) | Baseline, 6 months, 12 months, 18 months and 2 years
  Blood test at hospital or general practitioner
C-Reactive Protein (CRP) (intervention group) | Monthly until 2 years
  Blood test measured at home in a subgroup among the intervention group
Modified Health Assessment Questionnaire (MHAQ) | Baseline, 6 months, 12 months, 18 months, 2 years
  8 question concerning physical function, scored from 0 (no problems) to 3 (impossible to perform)
PROMIS Physical function | Baseline, 6 months, 12 months, 18 months, 2 years
  4 questions concerning physical function measured on a 5 point Likert scale
Pain (intervention group) | Baseline and monthly until 2 years
  Self-reported pain measured on a 11-point NRS (0=no pain; 10=worst possible pain)
Pain (control group) | Baseline, 6 months, 12 months, 18 months, 2 years
  Self-reported pain measured on a 11-point NRS (0=no pain; 10=worst possible pain)
Joint pain (intervention group) | Baseline and monthly until 2 years
  Self-reported joint pain measured on a 11-point NRS (0=no joint pain; 10=worst possible joint pain)
Joint pain (control group) | Baseline, 6 months, 12 months, 18 months, 2 years
  Self-reported joint pain measured on a 11-point NRS (0=no joint pain; 10=worst possible joint pain)
Sleep impairment | Baseline, 6 months, 12 months, 18 months, 2 years
  1 item from Pittsburgh Sleep Quality Index, self-reported sleep impairment in last month due to pain with 4 response categories ranging "Not during the past month" to "Three or more times a week" ; higher value indicate worse outcome.
Medication use | Baseline, 6 months, 12 months, 18 months, 2 years
  Medication, contomitant medication and any change in medication during the study period
Swollen joint count | Baseline, any hospital visits, 2 years
  Physician count of swollen joints; MCP 1-5, PIP 1-5, wrist, elbows, shoulders, ankles, MTP 1-5, at regular visits, extra visits, withdrawls, early discontinuation
Tender joint count | Baseline, any hospital visits, 2 years
  Physician count of tender joints; MCP 1-5, PIP 1-5, wrist, elbows, shoulders, ankles, MTP 1-5, at regular visits, extra visits, withdrawls, early discontinuation
Extra visits, telephone and video consultations | Through study completion, maximum 2 years
  Number of extra visits to the hospital or video consultations with a healthcare provider
Withdrawals/early discontinuation | Through study completion, maximum 2 years
  Number of withdrawals/early discontinuation
Physical activity | Baseline, 6 months, 12 months, 18 months, 2 years
  3 questions assessing frequency, intensity and duration of physical activity last week
Fatigue | Baseline, 6 months, 12 months, 18 months, 2 years
  Fatigue last week measured on an 11-point NRS (0=no fatigue, 10=worst possible fatigue)
Patient acceptable symptom state | Baseline, 6 months, 12 months, 18 months, 2 years
  one question assessing the patient acceptable symptom state last week, 5 response options from very good to very bad.
eHealth literacy | Baseline
  eHEALS questionnaire, 9 items measured on a 5 point Likert scale, with higher score indicating better health literacy
Patient-reported self-efficacy for using different digital devices, secure login and digital health services | Baseline
  Self-efficacy/confidence in using smartphone, tablet, computer, app's, secure login and digital health services. 6 items with Likert scale response categories: Never used, Very bad, Bad, Neither good nor bad, Good, Very good. Score range 1-5; higher scores indicate higher self-efficacy.
Patient satisfaction with care | Baseline, 6 months, 12 months, 18 months, 2 year
  1 item with five point response options ranging from "Very satisfied" to "Very dissatisfied", higher value indicate better outcome
Patient satisfaction with remote monitoring | 2 years
  Telehealth usability questionnaire (TUQ) 21 items scored from 1-7, higher score indicate higher satisfaction with telehealth

CONTACTS AND LOCATIONS:
Overall Officials: Anne Therese Tveter, PhD, Principal Investigator — Diakonhjemmet Hospital
Locations (1):
- Diakonhjemmet Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No
Data sharing of anonymous data may be possible upon reasonable request sent to the principal investigator.